CLINICAL TRIAL: NCT00143143
Title: Pregabalin BID Open-Label Add-On Trial: A Follow-Up Study To Determine Long-Term Safety and Efficacy in Patients With Partial Seizures
Brief Title: Pregabalin Open-Label Extension Trial in Patients With Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008-000-164
Record Dates: First submitted 2005-08-30; First posted 2005-09-02 (Estimated); Last update posted 2006-07-24 (Estimated); Status verified 2006-03

CONDITIONS: Epilepsies, Partial; Epilepsy, Complex Partial
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy, Complex Partial | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
The primary purpose of the protocol is to evaluate the long-term safety of pregabalin in patients with partial seizures.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met the inclusion criteria for Study 1008-157, have received double-blind study medication, and wish to receive open-label pregabalin
* Have the diagnosis of epilepsy with partial seizures and have a minimum of 4 partial seizures during the 6 weeks prior to screening
* Be currently taking 1 to 3 AEDs.

Exclusion Criteria:

* Have a treatable cause of seizures
* Experienced a serious adverse event during Study 1008-157 which was determined to be possibly related to study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-09; Study Completion 2006-02

PRIMARY OUTCOMES:
Safety assessments are performed at quarterly visits up until the study is closed.

SECONDARY OUTCOMES:
Seizure frequency is assessed throughout the study until the study is closed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- Austria (4):
  - Pfizer Investigational Site, Innsbruck
  - Pfizer Investigational Site, Mauer bei Amstetten
  - Pfizer Investigational Site, Sankt Pölten
  - Pfizer Investigational Site, Vienna
- Canada (8):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Barrie, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Trois-Rivières, Quebec
- France (9):
  - Pfizer Investigational Site, Marseille, Cedex 05
  - Pfizer Investigational Site, Paris, Cedex 13
  - Pfizer Investigational Site, Montpellier, Cedex 5
  - Pfizer Investigational Site, Lille, Cedex
  - Pfizer Investigational Site, Rennes, Cedex
  - Pfizer Investigational Site, Colomiers
  - Pfizer Investigational Site, Dommartin-lès-Toul
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Strasbourg
- Germany (10):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bielefeld
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Kehl
  - Pfizer Investigational Site, Marburg
  - Pfizer Investigational Site, Ulm
- Italy (4):
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Siena
- Pfizer Investigational Site, Vilnius, Lithuania
- Spain (4):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Girona, Gerona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Donostia / San Sebastian
- United Kingdom (3):
  - Pfizer Investigational Site, Glascow, Scotland
  - Pfizer Investigational Site, Fazakerley, Liverpool
  - Pfizer Investigational Site, York
- Pfizer Investigational Site